CLINICAL TRIAL: NCT02849899
Title: Prevention of New Onset Diabetes After Transplantation by a Short Term Treatment of Vildagliptin in the Early Post-transplant Period
Brief Title: Prevention of Diabetes After Transplantation by Vildagliptin in the Early Post-transplant Period
Acronym: PRODIG
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: University Hospital, Tours (Other); University Hospital, Lille (Other); Recherche Clinique Paris Descartes Necker Cochin Sainte Anne (Other); Amiens University Hospital (Other); University Hospital, Brest (Other); Rennes University Hospital (Other); Tenon Hospital, Paris (Other); Centre Hospitalier Universitaire de Nice (Other); University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: N/2015/70
Record Dates: First submitted 2016-07-19; First posted 2016-07-29 (Estimated); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Disorder Related to Renal Transplantation; Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Vildagliptin; Excipients

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vildagliptin (Active Comparator): Group 1 will be treated with Vildagliptin 50 or 100 mg/day for 2 months, then 25 or 50 mg/d for 1 month depending on their creatinine assay.
  Interventions: Drug: Vildagliptin
- Placebo (Placebo Comparator): Group 2 will be treated with placebo according to the same dosage.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vildagliptin — Galvus is prescribed as recommended by the marketing authorization. In adults, the recommended dose of Galvus is 100 mg per day (one tablet in the morning and another in the evening).
  In patients with moderate or severe kidney problems, the recommended dose is 50 mg once daily (one tablet in the morning).
  Patients with creatinine clearance greater than 50 ml/min the vildalgliptin dose will be 100 mg/day. For those whose clearance is less than 50 ml/min, the daily dose is 50 mg. The creatinine clearance will be measured each week.
  The treatment duration will be 3 months, divided into 2 months of complete treatment and one month of cessation treatment with half dose of vildagliptin.
  Other Names: Galvus
  Arms: Vildagliptin
Drug: Placebo — The placebo is the same as Galvus (packaging, shape, color, registration) but will contain only excipient. The given dose will also be identical.
  Other Names: Excipient
  Arms: Placebo

SUMMARY:
Post-transplant diabetes affects 15 to 20% of renal transplant patients and contributes to increased morbidity and reduced survival of transplants and patients. Corticosteroids, anti-calcineurin and mammilian Target OF Rapamycin (mTOR) inhibitors have a major diabetogenic impact and greatly contribute to the increase in diabetes prevalence after transplantation.

There are to date few studies concerning the pharmacological prevention of post-transplant diabetes. Hecking et al. have recently reported that a short treatment with insulin, administered immediately after transplantation, reduce the incidence of de novo diabetes one-year post-transplant. This study included 50 renal transplant patients and showed that a three months treatment of (Neutral Protamine Hagedorn) NPH insulin decreased HbA1c. The occurrence of diabetes, a secondary end-point, was reduced by 73% in the treated group.

No further pharmacological strategy has been developed to date. Relevant experimental evidences suggest that gliptins could be used in the pharmacological prevention of post-transplant diabetes. These drugs are inhibitors of dipeptidyl peptidase-4 (DPP-4), which inactivates the incretins, the glucagon-like peptide-1 (GLP-1) and the gastric inhibitory polypeptide (GIP). DPP-4 inhibition causes an increase in the GLP-1 and GIP concentrations which induce insulin secretion and inhibition of glucagon secretion. The gliptins are approved for the treatment of type 2 diabetes. Beyond the effects on blood glucose, gliptins have pleiotropic effects including a protective effect on β cells and anti-inflammatory effect.

The additional cost associated with new-onset diabetes after transplantation could be also significantly reduced by efficient prevention. A US study found that, for the period between 1994 and 1998, a newly diagnosed diabetic patient has cost $21,500 of medical expenses 2 years after transplantation. Moreover, transplantation resulting in one of the best increases of patients' quality of life, its estimate is essential in the treatment evaluation of this population.

ELIGIBILITY:
Inclusion Criteria:

* Major Patients (18 year old or older)
* Signature of informed consent
* Affiliation to a French social security or receiving such a scheme
* Patient receiving a first kidney transplant
* Patients considered at high risk of developing posttransplant diabetes having at least 2 of the 3 following criteria: Age> 50 years; BMI greater than 30 kg/m²; Direct Family history of type 2 diabetes
* Patients who can receive immunosuppressive therapy including tacrolimus, mycophenolic acid and steroids
* Patients in whom the cessation of steroids may be considered at the latest at Month 3 post-transplant

Exclusion Criteria:

* Legal disability or limited legal capacity
* Topic unlikely to cooperate in the study and / or low early cooperation by the investigator
* Patient without health insurance
* Pregnancy
* Patient in the period of exclusion of another study or under the "national register of volunteers."
* Inability to understand the reasons for the study; psychiatric disorders judged by the investigator to be incompatible with the inclusion in the study
* Active infection
* Infection with Hepatitis C virus
* A history of diabetes
* Multi-Organ Transplantation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2018-10-26 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Diabetes event | 1 year
  The primary endpoint is the proportion of diabetic patients 1 year after transplantation.
  Diabetic patients are defined as one of the following proposals:
  * Patients receiving a diabetic treatment
  * Patients have a fasting glucose above 7 mmol/l
  * Patients with an abnormal oral glucose tolerance test (OGTT)

SECONDARY OUTCOMES:
Glycemic control | 3, 6 and 12 months
  The criteria for secondary assessments are abnormal blood glucose measured by: the glycated hemoglobin (HbA1c) 3 months, 6 months and 12 months after transplantation.
Acute rejection, infections, graft and patient survival | 3, 6 and 12 months
  The occurrence of acute rejection, infection, graft loss and patient death 3 months, 6 months and 12 months after transplantation.
The health-related quality of life improvement | 3, 6 and 12 months
  The health-related quality of life (ReTRANSQOL questionnaire), 3 months, 6 months and 12 months after transplantation.
The cost-effectiveness ratio | 1 year
  The cost-effectiveness of prevention of diabetes with vildagliptin

CONTACTS AND LOCATIONS:
Overall Officials: Didier Ducloux, Pr., Principal Investigator — Besançon University Hospital, Nephrology department
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaiffe E, Crepin T, Bamoulid J, Courivaud C, Buchler M, Cassuto E, Albano L, Chemouny JM, Choukroun G, Hazzan M, Kessler L, Legendre C, Le Meur Y, Ouali N, Thierry A, Anota A, Nerich V, Limat S, Bonnetain F, Vernerey D, Ducloux D. PRODIG (Prevention of new onset diabetes after transplantation by a short term treatment of Vildagliptin in the early renal post-transplant period) study: study protocol for a randomized controlled study. Trials. 2019 Jun 21;20(1):375. doi: 10.1186/s13063-019-3392-6. PMID 31227028